CLINICAL TRIAL: NCT02251119
Title: The Pharmacodynamic/Pharmacokinetic Interaction of Tipranavir and Ritonavir With Loperamide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.55
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Loperamide

ARMS (2):
- TPV (Experimental): Administration of LOP on days 1, 9 and 22
  Administration of TPV on days 4-9
  Administration of TPV/RTV on days 12-22
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Loperamide
- RTV (Experimental): Administration of LOP on days 1, 9 and 22
  Administration of RTV on days 4-9
  Administration of TPV/RTV on days 12-22
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Loperamide

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Loperamide

SUMMARY:
The objective of the study was to determine if the co-administration of loperamide (LOP) with tipranavir (TPV), ritonavir (RTV), or TPV plus RTV (TPV/r) caused a clinically significant change in the respiratory response to carbon dioxide (CO2), defined as a 10% decrease in the area under the pharmacodynamic effect/time curve or at least a 25% decrease in at least one pharmacodynamic time point.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give written informed consent in accordance with institutional and federal guidelines and to comply with the investigational nature of the study and the related requirements
2. Healthy males or females between 18 and 60 years of age inclusive
3. A body mass index (BMI) between 18 and 35 kg/m2
4. Ability to perform a respiratory depression test
5. Ability to swallow numerous large capsules without difficulty
6. In the opinion of the investigator, a reasonable probability for completion of the study
7. Acceptable laboratory values that indicated adequate baseline organ function were required at the time of screening. Laboratory values were considered to be acceptable if their severity was ≤Grade 1 based on the AIDS Clinical Trials Group Division of AIDS (DAIDS) Grading Scale. All abnormal laboratory values >Grade 1 (e.g., creatinine phosphokinase, amylase, triglycerides) were subject to approval by the clinical monitor or designee
8. Acceptable medical history, physical examination, ECG, and chest x-ray were required prior to entering the study
9. Willingness to abstain from alcohol from Day -2 to Day 24. In addition, red wine must not have been ingested within 14 days prior to Day 1 (Visit 2)
10. Willingness to abstain from ingesting grapefruit, grapefruit juice, Seville oranges, St. John's Wort and Milk Thistle, within 14 days of Day 1 (Visit 2) and for the duration of the study
11. Willingness to abstain from ingesting garlic supplements, or methylxanthine containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 72 hours of pharmacokinetic (PK) sampling days (Day 1 [Visit 2], Day 9 [Visit 3], Day 21-22 [Visit 4])
12. Willingness to abstain from the use of tobacco products for the duration of the study
13. Nonsmoker
14. Urine drug screen negative for illegal nonprescription drugs
15. Negative HIV serology
16. Negative serology for hepatitis B surface antigen and hepatitis C

Exclusion Criteria:

1. Female subjects who were of reproductive potential who:

   * Had a positive serum β-human chorionic gonadotropin test at Visit 1, or
   * Had not been using a barrier contraceptive method for at least 3 months prior to Visit 2 (Day 1), or
   * Were not willing to use a reliable method of double-barrier contraception (such as a diaphragm with spermicidal cream/jelly or condoms with spermicidal foam) during the trial and 30 days after completion/termination of the trial, or
   * Were breast-feeding
2. Participation in another trial with an investigational medicine for 30 days prior to Day 1 (Visit 2)
3. Ingestion of any known enzyme-altering drug listed in the protocol 30 days prior to Day 1 (Visit 2)
4. Ingestion of grapefruit, grapefruit juice, St. John's Wort, Milk Thistle, Seville oranges and red wine within 14 days prior to Day 1 (Visit 2)
5. Ingestion of garlic supplements or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 72 hours of PK sampling days (Day 1 [Visit 2], Day 9 [Visit 3], Day 21-22 [Visit 4])
6. Ingestion of antibiotics within 10 days prior to Day 1 (Visit 2)
7. Inability to comply with investigator's instructions
8. History of gastrointestinal, hepatic, or renal disorders within 60 days of study entry
9. Recent or active alcohol abuse
10. Current use of tobacco products
11. Blood or plasma donations within 30 days prior to Day 1 (Visit 2)
12. Seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min
13. A history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering TPV or RTV or LOP to the subject
14. An acute illness within 2 weeks prior to Day 1 (Visit 2)
15. Current taking of any over-the-counter drug within 7 days prior to Day 1 (Visit 2) or current taking of any prescription drug that, in the opinion of the investigator in consultation with the clinical monitor and pharmacokineticist, might interfere with either the absorption, distribution or metabolism of the test substances
16. Hypersensitivity to TPV, RTV, or LOP
17. Administration of any antidiarrheal agent within 7 days of Day 1 (Visit 2)
18. Hypersensitivity to sulfonamide drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-07; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Maximum decrease in the percentage baseline CO2 response slope | up to 6 hours on days 1, 9 and 22
  rebreathing test
Zero-to-six hour area under the curve for the percentage baseline CO2 response slope profile | up to 6 hours on days 1, 9 and 22

SECONDARY OUTCOMES:
Change in the ratio between the diameter of the iris and pupil | Pupillary resonse to loperamide
  up to 6 hours on days 1, 9 and 22
Maximum plasma concentration | up to 75 h after drug administration
Minimum plasma concentration | up to 75 h after drug administration
Time to reach peak or maximum concentration | up to 75 h after drug administration
Terminal half life | up to 75 h after drug administration
Oral clearance | up to 75 h after drug administration
Area under the plasma concentration time curve | up to 75 h after drug administration
Number of subjects with adverse events | up to day 24